CLINICAL TRIAL: NCT07189806
Title: A Study of Mild, Moderate and Severe Asthma: Characterisation of Phenotypes and Endotypes and Longitudinal Associations With Exacerbations, Triggers and Disease Progression (MAPLE-UK)
Brief Title: Longitudinal Phenotyping and Endotyping Study in Adult Patients With Mild, Moderate, or Severe Asthma
Acronym: MAPLE-UK
Status: Recruiting | Type: Observational
Sponsor: Hvivo (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: HRD-AST-001
Record Dates: First submitted 2025-09-08; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Asthma (Diagnosis)
Keywords: Asthma; Severe; Moderate; Mild; Exacerbations; Longitudinal; Observational; Dyspnea; coughing; Inflammation; Bronchospasm
MeSH Terms: conditions — Asthma; Disease; Lymphoma, Follicular; Dyspnea; Cough; Inflammation; Bronchial Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood/Serum, Urine and Nasal samples:
  Some samples or portions of samples collected from participants may remain after the study is completed. Additionally, with written informed consent, extra optional blood samples may be collected.
  These leftover and/or additional samples and the clinical and research information that accompanies them may be useful for future research projects. If the participants consents, these remaining samples will become part of a collection to be stored at hVIVO's nominated laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and study aims:

The purpose of this research registry is to understand how asthma varies from person to person and monitor changes that may occur over time.

The effects that asthma has on the body will be assessed, by looking at different causes/triggers of flare-ups/exacerbations, asthma symptoms, and how inflammation of the airways may affect respiratory health over time.

The information obtained from this study will allow hVIVO to better understand respiratory disease progression and outcomes in asthma patients.

Who can participate:

Male or Female patients aged ≥ 18 years who are attending the hVIVO respiratory site clinics and have a clinical diagnosis of asthma.

What does the study involve:

The study will consist of a baseline clinic visit to confirm suitability and assess participants' asthma followed by approximately 5 annual clinic visits and follow-up phone calls, as necessary. Intermediate home self-assessments will also be scheduled for halfway between each annual clinic visit. Upon experiencing cold-like symptoms, participants will be asked to complete a at home self-nasal and throat swab as well as symptom, medication, and lung function home diary cards.

What are the possible benefits and risks of participating:

Taking part will not improve participants' health, although participants might benefit from a general health check at Screening as well as additional health checks and assessments of participants' inhaler technique during the conduct of the study.

There may be unexpected and unforeseen risks related to the study procedures. When attending for clinic visits, assessment will be performed by appropriately trained and qualified staff. Participants will be monitored for any procedure related symptoms such as, pain or bruising at the site where blood is drawn. Discomfort, sneezing, watery eyes, irritated nose, or nose bleeding during nasal sample collection. Light-headedness, dizziness, fatigue, coughing, shortness of breath, headaches, chest discomfort, throat irritation and itching during lung function testing. Skin irritation and allergic reactions from skin prick testing.

Should participants experience any of these symptoms, trained staff will be on hand to provide the appropriate medical treatment.

The Methacholine bronchial challenge test is also likely to cause asthma symptoms such as wheezing, shortness of breath, and chest tightness. In rare cases, the test can cause severe bronchospasm.

After the test or if the bronchospasm is severe, the technician will give the participant medication to inhale that will open the airways.

If the participant experiences any asthma exacerbation as a result of the methacholine test, the exacerbation management guidelines will be used to assess the participant and guide treatment.

Only participants that are not contraindicated for a methacholine test will have this performed.

For the at home assessments, participants will receive proper training on how to perform these during screening visit and as needed during each clinic follow-up visit.

Any abnormalities identified during the study will be communicated to the participant, as well as to the participant's GP or a specialist if necessary.

Where is the study run from:

hVIVO Services Limited - UK. Please see Participating Centres listed above for address.

When is the study starting and how long is it expected to run for:

The study began enrolling participants from 08th August 2025 and is unending, with an initial cohort of 235 expected to last approximately 5 years for each participant.

Who is funding the study:

hVIVO Services Limited

Who is the main contact:

Alex Mann - projectadmin@hvivo.com

DETAILED DESCRIPTION:
The MAPLE study is a prospective observational study of asthma patients at the hVIVO clinical site. This study is designed as a long-term research vehicle with no limit to enrolment or any time defined end.

The MAPLE study will enrol from across the spectrum of asthma severity and specifically include a strong representation of mild asthma, it will also include well controlled and less controlled, Type 2 high and low participants. Key aims will focus on the risk of progression and influence of various triggers, frequency of clinical and inflammatory risk factors (as and when participants progress from mild to more severe asthma), and assess variability and stability of respiratory and blood biomarkers and their ability to inform and predict risk (including inflammatory biomarkers, and blood cells).

An initial cohort of up to at least 235 asthma patients, ≥18 years of age who attend hVIVO's clinical site, are planned to be enrolled. Longer-term clinical outcomes will be monitored for at least 5 years.

Data will be collected both at yearly clinic visits as well as at planned intermediate at-home self-monitoring intervals.

The study design is divided into the following study phases:

1. Baseline: Participants who have shown an interest in hVIVO will be invited to a screening visit, where where details of the study will be provided. Historical generic screening data collected through the hVIVO generic screening process may be transferred to this study after the study-specific consent form has been signed by the participant.

   * Study Specific Informed consent: Volunteers deemed ineligible by the Investigator during the consenting consultation will be excluded and will not proceed. If eligible, the volunteer will continue to have the following assessments and procedures performed but, may be excluded at any point should any of the procedures listed below immediately demonstrate ineligibility.

     * Eligibility criteria
     * Demographics
     * Risk factor assessments: smoking status and history, occupational exposure to pollutants, allergens.
     * Socioeconomic status/income: employment status and Work Productivity and Activity Impairment Asthma Questionnaire (WPAI).
     * Height, weight, BMI, waist circumference
     * Medical & medication history, patient diagnosis, disease severity, age at diagnosis, personal and family history of asthma/COPD and allergies
     * Comorbidities (including associated medications)
     * Exacerbation history, asthma complications, respiratory diseases (e.g., RTI)
     * Asthma treatment(s) during previous 12 months - duration and posology, adherence, reasons for switching/discontinuation, satisfaction
     * Asthma medication assessment - inhaler technique & inhaler training if needed
     * Concomitant medications
     * Healthcare resource utilization
     * Urine drugs of misuse screen
     * Urinalysis
     * Alcohol breath test
     * Urine pregnancy test, if applicable
     * Complete physical examination
     * Vital signs (HR, RR, SBP, DBP, SpO2) and tympanic temperature
     * 12-lead ECG
     * Fractional exhaled nitric oxide Test (FeNO)
     * Forced Oscillation Technique (FOT)
     * Peak Flow Measurement (PEF) self-test
     * Spirometry (including PEF)
     * Symptom Diary Card
     * Home Participant Diary Card including: Symptom diary card, PEF (self-test), asthma medications, cold perception and night disturbances and Asthma questionnaires (ACQ-6).
     * Asthma Control Questionnaire (ACQ-7)
     * Asthma Impairment and Risk Questionnaire (AIRQ)
     * Quality of Life Questionnaire(s) e.g. Asthma Quality of Life (AQLQ)
     * Hematology
     * Biochemistry
     * Blood - biomarkers
     * Serum - humoral immunity & cytokine/chemokine markers
     * Whole blood for cell-mediated immunity
     * RNA PAXgene - transcriptomics
     * DNA PAXgene - genomics
     * Nasosorption - biomarkers
     * Nasopharyngeal swab - respiratory pathogen screen
     * Exhaled breath sampling method(s) (e.g. exhaled breath condensate)
     * Induced sputum - cells, transcriptomics and biomarkers.
     * Allergen skin prick test
     * Methacholine challenge (AHR)
     * Bronchodilator responsiveness

   For participants enrolled in to Optional Sub-studies, the following additional assessments may be performed at the screening visit and at any time on and between annual clinic visits and may occur once or more for consented participants throughout the study.
   * Physiological measurement devices to measure parameters such as vital signs, sleep, cough
   * Nasal Allergy challenge (NAC)
   * Bronchial Allergen challenge (BAC)
   * Viral challenge e.g. rhinovirus
2. Follow-up Phase including Intermittent at home assessments:

Participants will attend yearly clinic follow-up visits and will be required to complete at home self-assessments at 6 monthly intervals and when experiencing symptoms of a respiratory infection.

During each yearly clinic visit, procedures similar to the baseline visit will be performed as appropriate to reassess change in participants' asthma and medications.

Interim at home assessments will include:

* Home Participants Diary Card that includes assessments of:

  * Symptoms
  * Asthma medication usage
  * Peak expiratory flow (PEF)
  * Cold perception
  * Night disturbances
  * Asthma Control Questionnaire (ACQ-6).
  * Exacerbation history
* Collection of respiratory samples (self-sampling) when experiencing cold-like symptoms.

Participants may withdraw from the study at any time, and all efforts will be made to document any reasons for withdrawal and to complete required end-of-study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged ≥ 18 years and older who have signed an Informed Consent form.
2. All patients who attend the hVIVO respiratory site clinics who have a clinical diagnosis of asthma/any of the following:

   * Positive response to methacholine challenge test (AHR), or
   * Positive response to a bronchodilator responsiveness test, or
   * Peak Flow variability (i.e. highest - lowest PEF over the day/mean value of the two, × 100) > 20%, or
   * Documented response (defined as ΔFEV1 ≥ 12% and ≥ 200 mL) after a cycle (e.g., 4 weeks) of regular maintenance anti-asthma treatment, or
   * physician diagnosis of current asthma.
3. In the PI/investigator(s) opinion, will be able to follow the study requirements.

Exclusion Criteria:

1. Asthma patients who are not attending hVIVO respiratory site clinics.
2. Patients whose primary respiratory diagnosis (i.e. the condition causing most of their respiratory symptoms) is not asthma (however, a co-diagnosis of another respiratory disease such as COPD, bronchiectasis or interstitial lung disease together with asthma will be accepted)
3. Females who:

   1. Are breastfeeding, or
   2. Have a positive pregnancy test at any point during screening
4. Patients who, in the opinion of the physician, are unlikely to complete the 5 years of follow-up, e.g. poor literacy, substance abuse, life threatening comorbidities.
5. Contraindications for lung function testing, e.g., hemoptysis of unknown origin, history of pulmonary hypertension, previous pneumothorax, unstable cardiovascular status (severe heart failure, or ischemic heart disease), aneurysms (thoracic, abdominal or cerebral), recent eye surgery (e.g., cataract), recent thoracic or abdominal surgery.
6. Patients with lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend the hVIVO respiratory site clinics who have a clinical diagnosis and meet the inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2050-08-08 (Estimated); Study Completion 2050-08-08 (Estimated)

PRIMARY OUTCOMES:
Exacerbation history (number and severity) | Baseline, Year 1, 2, 3, 4, 5
  Medical review
Spirometry - change in Forced Expiratory Volume in 1 second (FEV1) (Litres [L]) | Change from baseline FEV1 at Year 1, 2, 3, 4, 5
  Lung function test
Spirometry - change in Forced Vital Capacity (FVC) (L) | Change from baseline FVC at Year 1, 2, 3, 4, 5
  Lung function test
Spirometry - change in Peak Expiratory Flow (PEF) (Litre/second [L/s]) | Change from baseline PEF at Year 1, 2, 3, 4, 5
  Lung function test
Spirometry - change in Forced Expiratory Flow at 25-75% of the forced vital capacity (FEF25-75%) (L/s) | Change from baseline FEF25-75% at Year 1, 2, 3, 4, 5
  Lung function test
Post-bronchodilator spirometry - FEV1 (L) | Optionally Year 1,2,3,4,5
  Bronchodilator responsiveness test
Post-bronchodilator spirometry - FVC (L) | Time Frame: Optionally Year 1,2,3,4,5
  Bronchodilator responsiveness test
Post-bronchodilator spirometry - PEF (L/s) | Optionally Year 1,2,3,4,5
  Bronchodilator responsiveness test
Post-bronchodilator spirometry - FEF25-75% (L/s) | Optionally Year 1,2,3,4,5
  Bronchodilator responsiveness test
Oscillometry - Absolute and change in R5-R20 kPa/L | Grouping, absolute and Change from baseline R5-R20 at Year 1, 2, 3, 4, 5
  Small airway test
Oscillometry - Absolute and change in AX kPa/L | Grouping, absolute and Change from baseline AX at Year 1, 2, 3, 4, 5
  Small Airway Test
Oscillometry - Absolute and change in X5 kPa/L | Grouping, absolute and Change from baseline X5 at Year 1, 2, 3, 4, 5
  Small Airway Test
Skin Prick Test - Qualitative atopy | Baseline, & optionally Year 1,2,3,4,5
  Atopy Test
Methacholine Test - provocative concentration (PC20) causing a 20% fall in (FEV1) (mg/mL) | Baseline, & optionally Year 1,2,3,4,5
  Airway Hyperreactivity Test
Fractional exhaled nitric oxide (FeNO) (parts per billion [ppb]) | Baseline, & Year 1,2,3,4,5
  Test to measure fractional exhaled nitric oxide (ppb) levels in exhaled breath
Absolute and change from baseline symptoms/symptom control assessed by the Asthma Control Questionnaire (ACQ®) | Baseline and Change from baseline ACQ mean scores at Year 1, 2, 3, 4, 5, & ad-hoc timepoints
  Patient reported outcome questionnaire
Absolute and change from baseline symptoms/symptom control assessed by the Asthma Impairment and Risk Questionnaire (AIRQ®) | Baseline and Change from baseline AIRQ scores at Year 1, 2, 3, 4, 5
  Patient reported outcome questionnaire
Absolute and change from baseline symptoms/symptom control assessed by the Asthma Quality of Life Questionnaire (AQLQ®) | Baseline and Change from baseline AQLQ scores optionally at Year 1, 2, 3, 4, 5
  Patient reported outcome questionnaire
Absolute and change from baseline symptoms assessed by self-reported ordinal scale diary card | Baseline and Change from baseline scores at Year 1, 2, 3, 4, 5, & ad-hoc timepoints
  Patient reported outcome questionnaire
Absolute and change from baseline symptoms assessed by self-reported visual analogue scale diary card | Baseline and Change from baseline scores at Year 1, 2, 3, 4, 5, & ad-hoc timepoints
  Patient reported outcome questionnaire
Patient reported cold perception | Baseline and Year 1, 2, 3, 4, 5, & ad-hoc timepoints
  Patient reported outcome questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lima, MD-PhD, Principal Investigator — Hvivo
Locations (1):
- hVIVO Services Limited, 40 Bank Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No